CLINICAL TRIAL: NCT04310787
Title: The Investigation on Long-term Outcomes and Prognostic Factors of Patients With Hepatitis B Related Acute-on-chronic Liver Failure
Brief Title: Long-term Prognosis of Patients With Hepatitis B Related Acute-on-chronic Liver Failure
Status: Recruiting | Type: Observational
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professer, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: PL12
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Hepatitis B; Acute-On-Chronic Liver Failure
Keywords: Hepatitis B; Acute-On-Chronic Liver Failure; Prognosis
MeSH Terms: conditions — Hepatitis B; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HBV-ACLF: To investigate the clinical events and prognosis of patients with hepatitis b associated acute on-chronic liver failure

SUMMARY:
This study is to investigate the long-term outcomes and prognostic risk factors in patients recovered from hepatitis B virus related acute on-chronic liver failure.

DETAILED DESCRIPTION:
Chronic acute liver failure (ACLF) is a systemic multi-organ failure driven by acute liver injury in the basis of chronic liver disease. The main cause of chronic acute liver failure in China is hepatitis b virus infection.Previous studies on the prognosis of acute on-chronic liver failure mainly focused on the short-term survival rate and the follow-up time was relatively short, while the study on the long-term prognosis of patients with spontaneous recovery of chronic acute liver failure was still lack-ing. Thus,this study mainly retrospectively analyzed the clinical data of patients with chronic hepatitis b related acute liver failure admitted to the department of infectious diseases, the third affiliated hospital of sun yat-sen university, and con-ducted telephone follow-up survey to analyze the long-term prognosis of patients with chronic hepatitis b related acute on-chronic liver failure.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years old;
* The diagnosis consistent with hepatitis b associated chronic acute liver failure；
* After hospitalization, the survival time > 90 days；
* The inpatient clinical data are complete.

Exclusion Criteria:

* Human immunodeficiency virus infection or congenital immune deficiency diseases;
* Liver cancer and other tumors, autoimmune liver disease, genetic and metabolic liver disease, or other serious diseases that significantly affect patient survival;
* Other conditions that the researchers judged not appropriate for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study population were patients with hepatitis b-related acute on-chronic liver failure in the department of infectious diseases, the third affiliated hospital of sun yat-sen university.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
adverse events | 5 years
  Adverse events included decompensated cirrhosis, hepatocellular carcinoma, liver transplantation, and death.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in this article (text, tables, figures and appendices) will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be shared beginning 3 months and ending 5 years following the article publication.
Access Criteria: Proposals should be directed to xxx@yyy. To gain access, data requestors need to sign a data access agreement.